CLINICAL TRIAL: NCT05516303
Title: Pharmacogenetic Investigation of Susceptibility to Liver Toxicity in Patients With Multiple Sclerosis Treated With Fingolimod
Brief Title: Pharmacogenetics of Liver Toxicity in Patients With Multiple Sclerosis Treated With Fingolimod
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0041
Record Dates: First submitted 2022-06-10; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
Keywords: Fingolimod; hepatic adverse events; polymorphism
MeSH Terms: conditions — Multiple Sclerosis | interventions — Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: MS patients treated with fingolimod who experienced liver enzymes elevation
  Interventions: Genetic: Genetic polymorphism; Diagnostic Test: Measurement of fingolimod and fingolimod-phosphate concentrations
- Control: MS patients treated with fingolimod not experiencing elevated liver enzymes
  Interventions: Genetic: Genetic polymorphism; Diagnostic Test: Measurement of fingolimod and fingolimod-phosphate concentrations

INTERVENTIONS:
Genetic: Genetic polymorphism — One blood tube will be taken for genetic testing
Diagnostic Test: Measurement of fingolimod and fingolimod-phosphate concentrations — Measurement of fingolimod and fingolimod-phosphate concentrations before usual drug administration time

SUMMARY:
To investigate whether polymorphic differences can be identified between Multiple Sclerosis patients developing elevated liver enzymes (defined as ALT, AST, GGT or bilirubinemia levels five above the upper normal limit on at least one) compared to those not developing elevated liver enzymes after exposure to fingolimod for multiple sclerosis.

DETAILED DESCRIPTION:
PURPOSE: To investigate whether polymorphic differences can be identified between Multiple sclerosis (MS) patients treated by fingolimod who had liver enzymes elevation compared to those who do not.

OBJECTIVE: To determine whether elevated liver enzyme tests (ALT, AST, GGT or bilirubinemia above the upper limit of normal) in MS patients treated with fingolimod is associated with genetic polymorphisms.

METHOD OF RECRUITMENT:

Patients will be identified through a clinic database and chart reviews. A phone call will be made to determine interest. Upon a follow-up neurological consultation, consent into study will be sought.

PROCEDURES:

Blood samples will be collected for genetic analyses, fingolimod and fingolimod-phosphate quantification and a questionnaire will be administered

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years)
* Have a definite Multiple Sclerosis with a relapsing-remitting course (McDonald criteria)
* Treated with fingolimod
* Have given consent and signed an informed consent form

Exclusion Criteria:

* an elevated liver test result on baseline before starting fingolimod treatment
* presence of a viral, hereditary or auto-immune liver pathology
* Time of fingolimod exposure lower than three months
* Woman currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis (MS) patients attending out-patient neurological consultations in Caen University Hospital, with a relapsing-remitting disease course, and prescribed fingolimod as a disease-modifying drug for MS.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
CYP4F2 polymorphism frequency in case and control groups | At inclusion
  Proportion of CYP4F2 polymorphism in case and control groups

SECONDARY OUTCOMES:
Fingolimod concentrations in case and control groups | At inclusion
  Trough concentration of fingolimod in blood samples determined by liquid chromatography-tandem mass spectrometry (LC-MS)
Fingolimod-phosphate concentrations in case and control groups | At inclusion
  Trough concentration of fingolimod-phosphate in blood samples determined by liquid chromatography-tandem mass spectrometry (LC-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Defer, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided